CLINICAL TRIAL: NCT04992468
Title: Dual Trigger vs.GnRH-a Trigger for Elective Fertility Preservation. A Randomized Controlled Trial
Brief Title: Dual Trigger for Elective Fertility Preservation
Acronym: DUAL-T
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación Santiago Dexeus Font (Other)
Responsible Party: Sponsor
Organization: Fundacion Dexeus (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FSD-PSE-2021-09; 2021-002467-22 (EudraCT Number)
Record Dates: First submitted 2021-07-05; First posted 2021-08-05 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GnRH-a+rhCG (Experimental): Ovulation triggering with GnRH-a+rhCG
  Interventions: Drug: Ovulation triggering with GnRH-a+rhCG
- GnRH-a (Active Comparator): Ovulation triggering with GnRH-a
  Interventions: Drug: Ovulation triggering with GnRH-a

INTERVENTIONS:
Drug: Ovulation triggering with GnRH-a+rhCG — recombinant follicle stimulating hormone (rFSH) 225-300 IU (Gonal-F®/Puregon®/ Ovaleap®/Rekovelle®) Micronized progesterone 200mg (Utrogestan®) Ovulation trigger: Triptorelin 0.2 mg (Decapeptyl®) + Recombinant human chorionic gonadotropin (rhCG) 250μg (Ovitrelle®)
  Arms: GnRH-a+rhCG
Drug: Ovulation triggering with GnRH-a — rFSH 225-300 IU (Gonal-F®/Puregon®/Ovaleap®/ Rekovelle®) Micronized progesterone 200mg (Utrogestan®) Ovulation trigger: Triptorelin 0.2 mg (Decapeptyl®)
  Arms: GnRH-a

SUMMARY:
The widespread availability of efficient contraception as well as women's increased education has led to childbearing postponement. Combined with the increased recognition of the concept of "ovarian aging", this has opened the Pandora´s box of EOC, which is currently considered a safe and cost-efficient approach among assisted reproduction techniques.

Previous studies have shown that two main factors determine the CLBR after EOC: 1) patient's age at the time of oocyte banking, and 2) the number of oocytes retrieved. Therefore, measures aiming at increasing the oocyte yield, specially the number of mature oocytes retrieved, will maximize the success of this technique.

In the last few years, the dual trigger for final oocyte maturation has emerged has an approach that seems to improve both oocyte yield and quality when compared to the hCG trigger alone. Nowadays, the standard of care in EOC patients is final oocyte maturation with a single bolus of GnRH-a. Understanding the impact of the dual trigger on the number of MII oocytes retrieved in patients undergoing EOC will improve the treatment protocols and allow for a better patient counselling.

DETAILED DESCRIPTION:
Elective oocyte cryopreservation (EOC) has been gaining increasing importance in the last few years, driven by the widespread information regarding the concept of 'age-related fertility decline', as well as the availability of efficient contraception and women's increasing educational and professional aspirations. Considering the similar clinical outcomes regarding live birth rate after vitrified-warmed and fresh oocytes and the proven cost-effectiveness of this approach, oocyte banking is now considered an efficient technique in assisted reproduction.

Previous studies have shown that both patient's age and the number of oocytes retrieved have a significant impact on the cumulative live birth rate (CLBR) in patients undergoing EOC, highlighting the importance of maximizing oocyte yield in these patients.

In all these former reports, final follicular maturation was triggered by one bolus of human chorionic gonadotropin (hCG) or, following recent trends in clinical practice, by a single bolus of Gonadotropin Releasing Hormone agonist (GnRH-a).

More recently, the concomitant administration of both GnRH-a and a bolus of HCG prior to oocyte retrieval (dual trigger) has been proposed as a new strategy for final follicular maturation, aiming to improve oocyte and embryo quality . When compared to HCG trigger, the dual trigger adds the more physiologic follicular stimulating hormone (FSH) and luteinizing hormone (LH) peak provided by GnRH-a. With this approach, several studies have reported an increase in the number of MII oocytes retrieved, as well as in the number of good quality embryos and improved pregnancy outcomes in different subpopulations of infertile patients.

Nowadays, the standard of care in patients undergoing a freeze-all approach, either for oocyte or embryo cryopreservation, is final follicular maturation with GnRH-a due to its more physiologic and shorter surge of both LH and FSH, terminating 24h after its onset, and reducing the risk of ovarian hyperstimulation syndrome (OHSS). So far, no study has compared the dual trigger approach to the use of a single bolus of GnRH-a. By adding HCG activity and, therefore, generating higher intracellular cyclic adenosine monophosphate (cAMP) accumulation, an amplification of the steroidogenic response of the pre-ovulatory follicle might be achieved with the dual trigger when compared to the GnRH-a trigger alone.

Therefore, the investigators set out to perform this randomized controlled trial aiming to compare, for the first time, the dual trigger and the GnRH-a trigger regarding the number of MII oocytes retrieved in patients undergoing EOC.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to sign the Patient Consent Form and adhere to study visitation schedule
* antral follicle count (AFC) <20
* Anti-Mullerian hormone (AMH) ≤3ng/ml (AMH result of up to one year will be valid)
* Age >=18 and ≤40 years
* BMI >18 and <30 kg/m2

Exclusion Criteria:

* Medically indicated fertility preservation
* AFC ≥ 20
* Polycystic ovarian syndrome (PCOS) according to the Rotterdam criteria
* FSH ≥ 20
* History of untreated autoimmune, endocrine or metabolic disorders
* Contraindication for hormonal treatment
* Recent history of severe disease requiring regular treatment (clinically significant concurrent medical condition that could compromise subject safety or interfered with the trial assessment).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 136 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2023-04-25 (Actual)

PRIMARY OUTCOMES:
Number of mature oocytes (MIIs) retrieved | 7 -20 days from initiation of ovarian stimulation

SECONDARY OUTCOMES:
Number of oocytes retrieved | 7 -20 days from initiation of ovarian stimulation
Change in Progesterone values | Day 1 of ovarian stimulation, Day of HCG/HCG+Decapeptyl administration and Day after HCG/HCG+Decapeptyl
Change in Estradiol values | Day 1 of ovarian stimulation, Day of HCG/HCG+Decapeptyl administration and Day after HCG/HCG+Decapeptyl
Change in FSH values | Day 1 of ovarian stimulation, Day of HCG/HCG+Decapeptyl administration and Day after HCG/HCG+Decapeptyl
Change in LH values | Day 1 of ovarian stimulation, Day of HCG/HCG+Decapeptyl administration and Day after HCG/HCG+Decapeptyl
Ovarian hyperstimulation syndrome (OHSS) (percent) | Until 15 days after the end of ovarian stimulation

OTHER OUTCOMES:
Incidence of adverse events and serious adverse events | Until 15 days after the end of ovarian stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos P Polyzos, MD PhD, Study Chair — Hospital Universitari Dexeus; Ana Neves, MD, Principal Investigator — Hospital Universitari Dexeus
Locations (1):
- Hospital Universitario Quiron Dexeus, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ovarian Stimulation TEGGO, Bosch E, Broer S, Griesinger G, Grynberg M, Humaidan P, Kolibianakis E, Kunicki M, La Marca A, Lainas G, Le Clef N, Massin N, Mastenbroek S, Polyzos N, Sunkara SK, Timeva T, Toyli M, Urbancsek J, Vermeulen N, Broekmans F. ESHRE guideline: ovarian stimulation for IVF/ICSIdagger. Hum Reprod Open. 2020 May 1;2020(2):hoaa009. doi: 10.1093/hropen/hoaa009. eCollection 2020. PMID 32395637
- [Background] Casarini L, Lispi M, Longobardi S, Milosa F, La Marca A, Tagliasacchi D, Pignatti E, Simoni M. LH and hCG action on the same receptor results in quantitatively and qualitatively different intracellular signalling. PLoS One. 2012;7(10):e46682. doi: 10.1371/journal.pone.0046682. Epub 2012 Oct 5. PMID 23071612
- [Background] Cobo A, Garcia-Velasco J, Domingo J, Pellicer A, Remohi J. Elective and Onco-fertility preservation: factors related to IVF outcomes. Hum Reprod. 2018 Dec 1;33(12):2222-2231. doi: 10.1093/humrep/dey321. PMID 30383235
- [Background] Cobo A, Garcia-Velasco JA, Coello A, Domingo J, Pellicer A, Remohi J. Oocyte vitrification as an efficient option for elective fertility preservation. Fertil Steril. 2016 Mar;105(3):755-764.e8. doi: 10.1016/j.fertnstert.2015.11.027. Epub 2015 Dec 10. PMID 26688429
- [Background] Devine K, Mumford SL, Goldman KN, Hodes-Wertz B, Druckenmiller S, Propst AM, Noyes N. Baby budgeting: oocyte cryopreservation in women delaying reproduction can reduce cost per live birth. Fertil Steril. 2015 Jun;103(6):1446-53.e1-2. doi: 10.1016/j.fertnstert.2015.02.029. Epub 2015 Mar 23. PMID 25813281
- [Background] Ding N, Liu X, Jian Q, Liang Z, Wang F. Dual trigger of final oocyte maturation with a combination of GnRH agonist and hCG versus a hCG alone trigger in GnRH antagonist cycle for in vitro fertilization: A Systematic Review and Meta-analysis. Eur J Obstet Gynecol Reprod Biol. 2017 Nov;218:92-98. doi: 10.1016/j.ejogrb.2017.09.004. Epub 2017 Sep 14. PMID 28957685
- [Background] Doyle JO, Richter KS, Lim J, Stillman RJ, Graham JR, Tucker MJ. Successful elective and medically indicated oocyte vitrification and warming for autologous in vitro fertilization, with predicted birth probabilities for fertility preservation according to number of cryopreserved oocytes and age at retrieval. Fertil Steril. 2016 Feb;105(2):459-66.e2. doi: 10.1016/j.fertnstert.2015.10.026. Epub 2015 Nov 18. PMID 26604065
- [Background] Fauser BC, de Jong D, Olivennes F, Wramsby H, Tay C, Itskovitz-Eldor J, van Hooren HG. Endocrine profiles after triggering of final oocyte maturation with GnRH agonist after cotreatment with the GnRH antagonist ganirelix during ovarian hyperstimulation for in vitro fertilization. J Clin Endocrinol Metab. 2002 Feb;87(2):709-15. doi: 10.1210/jcem.87.2.8197. PMID 11836309
- [Background] Golan A, Weissman A. Symposium: Update on prediction and management of OHSS. A modern classification of OHSS. Reprod Biomed Online. 2009 Jul;19(1):28-32. doi: 10.1016/s1472-6483(10)60042-9. PMID 19573287
- [Background] Goldman RH, Racowsky C, Farland LV, Munne S, Ribustello L, Fox JH. Predicting the likelihood of live birth for elective oocyte cryopreservation: a counseling tool for physicians and patients. Hum Reprod. 2017 Apr 1;32(4):853-859. doi: 10.1093/humrep/dex008. PMID 28166330
- [Background] Griffin D, Feinn R, Engmann L, Nulsen J, Budinetz T, Benadiva C. Dual trigger with gonadotropin-releasing hormone agonist and standard dose human chorionic gonadotropin to improve oocyte maturity rates. Fertil Steril. 2014 Aug;102(2):405-9. doi: 10.1016/j.fertnstert.2014.04.028. Epub 2014 May 17. PMID 24842671
- [Background] Haas J, Bassil R, Samara N, Zilberberg E, Mehta C, Orvieto R, Casper RF. GnRH agonist and hCG (dual trigger) versus hCG trigger for final follicular maturation: a double-blinded, randomized controlled study. Hum Reprod. 2020 Jul 1;35(7):1648-1654. doi: 10.1093/humrep/deaa107. PMID 32563188
- [Background] Lin MH, Wu FS, Lee RK, Li SH, Lin SY, Hwu YM. Dual trigger with combination of gonadotropin-releasing hormone agonist and human chorionic gonadotropin significantly improves the live-birth rate for normal responders in GnRH-antagonist cycles. Fertil Steril. 2013 Nov;100(5):1296-302. doi: 10.1016/j.fertnstert.2013.07.1976. Epub 2013 Aug 28. PMID 23993928
- [Background] van Loendersloot LL, Moolenaar LM, Mol BW, Repping S, van der Veen F, Goddijn M. Expanding reproductive lifespan: a cost-effectiveness study on oocyte freezing. Hum Reprod. 2011 Nov;26(11):3054-60. doi: 10.1093/humrep/der284. Epub 2011 Sep 6. PMID 21896545
- [Background] Mills M, Rindfuss RR, McDonald P, te Velde E; ESHRE Reproduction and Society Task Force. Why do people postpone parenthood? Reasons and social policy incentives. Hum Reprod Update. 2011 Nov-Dec;17(6):848-60. doi: 10.1093/humupd/dmr026. Epub 2011 Jun 7. PMID 21652599
- [Background] Montoya-Botero P, Martinez F, Rodriguez-Purata J, Rodriguez I, Coroleu B, Polyzos NP. The effect of type of oral contraceptive pill and duration of use on fresh and cumulative live birth rates in IVF/ICSI cycles. Hum Reprod. 2020 Apr 28;35(4):826-836. doi: 10.1093/humrep/dez299. PMID 32163564
- [Background] Orvieto R. Triggering final follicular maturation: hCG, GnRH-agonist, or both, when and to whom? J Assist Reprod Genet. 2017 Sep;34(9):1231-1232. doi: 10.1007/s10815-017-0982-7. Epub 2017 Jun 27. No abstract available. PMID 28656537
- [Background] Youssef MA, Van der Veen F, Al-Inany HG, Mochtar MH, Griesinger G, Nagi Mohesen M, Aboulfoutouh I, van Wely M. Gonadotropin-releasing hormone agonist versus HCG for oocyte triggering in antagonist-assisted reproductive technology. Cochrane Database Syst Rev. 2014 Oct 31;2014(10):CD008046. doi: 10.1002/14651858.CD008046.pub4. PMID 25358904
- See also: Department of Obstetrics, Gynaecology and Reproduction Hospital Universitari Quiron Dexeus — http://www.dexeus.com